CLINICAL TRIAL: NCT05422313
Title: Assessment of Galectin-9 in Rheumatoid Arthritis and Its Correlation With Disease Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan mostafa Mohamed Abdelal, principle investigator, Assiut University
Other Study IDs: VDSF
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 56 patients with RA.: Patients age is > 20 years old.
- : 30 age-matched Healthy: Individual must be without a prior history of chronic inflammation or any form of arthritis. - .

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease in which a symmetrical Synovial inflammation, bone destruction occur in both small and big Joints. If left untreated, this illness does not generally cause death, but it does drastically affect the quality of life and life expectancy of patients. Although there is no cure for RA, patients are generally on long-term long-acting disease-modifying anti-rheumatic medications (DMARDs) to control joint inflammation, reduce joint damage, maintain joint function, and keep the illness in remission.

RA disease activity could be detected be DAS28 score. The DAS28 is a four-item scale that gives an absolute number reflecting disease activity. It includes the number of swollen and tender joints (SJC, TJC), the visual analogue scale of patients' assessment of their general health (VAS-GH), and the erythrocyte sedimentation rate (ESR) in the first hour.

In the pathophysiology of RA, cytokine networks play a crucial role. Rheumatoid inflammation has been linked to the generation of proinflammatory cytokines throughout time. Increased cytokine levels, such as tumour necrosis factor (TNF) and interleukin-6 (IL-6), represent rheumatoid synovial inflammation and have been linked to RA disease activity and anti-cytokine therapeutic response. The relationship between circulating cytokine levels and the phenotype of RA illness is, however, poorly understood.

Anti-citrullinated peptide antibodies (ACPA) are effective in the diagnosis of RA and have been linked to joint destruction progression and therapy response in RA patients. However, the relationship between ACPA status and proinflammatory cytokines during the course of RA illness is yet unknown.

Galectins are lectins with carbohydrate recognition domains (CRDs) that are extremely similar in sequence and exclusively bind to β--galactoside carbs. There are at least 15 galectins found in mammals, each having one or two CRDs comprising roughly 130 amino acids. Galectins have a wide range of activities due to their ubiquitous distribution, including mRNA splicing, programmed cell death, cell cycle control, activation, adhesion, migration, and cell differentiation.

Galectin-9 (Gal-9) is abundantly present in lymph nodes, bone marrow, liver, thymus, and spleen. It is expressed by immune cells, endothelial cells, and fibroblasts and plays an important role in regulating inflammation and immune reactions. Gal-9 is a ligand for T cell immunoglobulin and mucin-containing-moleculte-3 (Tim-3) that is expressed on CD4+ T helper (Th) 1 and Th17 and sends inhibitory signals to Tim-3. As a result of its interaction with Tim-3, Gal-9 suppresses pro-inflammatory T cell responses, and the Gal-9/Tim-3 pathway causes apoptosis of CD4+ Th1 or Th17 cells.

Considering that RA is a Th1-polarized autoimmune illness, dysregulated Gal-9 levels may induce an innate/adaptive immunity imbalance, resulting in pathological rheumatoid inflammation. Gal-9 has been demonstrated to mediate angiogenesis and inflammatory cell infiltration in inflammatory arthritis.

These findings show that Gal-9 may have a role in the inflammatory processes of rheumatoid arthritis. As a result, we concentrated on Gal-9 and postulated that it could be involved in the pathogenesis of RA. The levels of serum Gal-9 in individuals with RA were studied in this study, and the results were compared to clinical indicators

ELIGIBILITY:
Inclusion Criteria:

* Patients age is > 20 years old.
* All rheumatoid arthritis patients must fulfill the 2010 ACR/EULAR criteria for RA.

Exclusion Criteria:

* Patients age is < 20 years old.
* Patient with evidence of any concomitant inflammatory disease, Acute infection or chronic inflammatory status.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalized patients
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
To correlate galectin-9 level with RA disease activity. | 1.5 years
  use galectin-9 to determine disease activity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Floudas A, Canavan M, McGarry T, Mullan R, Nagpal S, Veale DJ, Fearon U. ACPA Status Correlates with Differential Immune Profile in Patients with Rheumatoid Arthritis. Cells. 2021 Mar 14;10(3):647. doi: 10.3390/cells10030647. PMID 33799480
- [Background] Gieseke F, Kruchen A, Tzaribachev N, Bentzien F, Dominici M, Muller I. Proinflammatory stimuli induce galectin-9 in human mesenchymal stromal cells to suppress T-cell proliferation. Eur J Immunol. 2013 Oct;43(10):2741-9. doi: 10.1002/eji.201343335. Epub 2013 Jul 23. PMID 23817958
- [Background] Golden-Mason L, McMahan RH, Strong M, Reisdorph R, Mahaffey S, Palmer BE, Cheng L, Kulesza C, Hirashima M, Niki T, Rosen HR. Galectin-9 functionally impairs natural killer cells in humans and mice. J Virol. 2013 May;87(9):4835-45. doi: 10.1128/JVI.01085-12. Epub 2013 Feb 13. PMID 23408620
- [Background] Yap HY, Tee SZ, Wong MM, Chow SK, Peh SC, Teow SY. Pathogenic Role of Immune Cells in Rheumatoid Arthritis: Implications in Clinical Treatment and Biomarker Development. Cells. 2018 Oct 9;7(10):161. doi: 10.3390/cells7100161. PMID 30304822
- [Background] McInnes IB, Schett G. Cytokines in the pathogenesis of rheumatoid arthritis. Nat Rev Immunol. 2007 Jun;7(6):429-42. doi: 10.1038/nri2094. PMID 17525752
- [Background] Naranjo A, Ojeda S, Francisco F, Erausquin C, Rua-Figueroa I, Rodriguez-Lozano C. Fibromyalgia in patients with rheumatoid arthritis is associated with higher scores of disability. Ann Rheum Dis. 2002 Jul;61(7):660-1. doi: 10.1136/ard.61.7.660. No abstract available. PMID 12079919
- [Background] Ogata A, Kato Y, Higa S, Yoshizaki K. IL-6 inhibitor for the treatment of rheumatoid arthritis: A comprehensive review. Mod Rheumatol. 2019 Mar;29(2):258-267. doi: 10.1080/14397595.2018.1546357. Epub 2019 Jan 3. PMID 30427250
- [Background] O'Brien MJ, Shu Q, Stinson WA, Tsou PS, Ruth JH, Isozaki T, Campbell PL, Ohara RA, Koch AE, Fox DA, Amin MA. A unique role for galectin-9 in angiogenesis and inflammatory arthritis. Arthritis Res Ther. 2018 Feb 12;20(1):31. doi: 10.1186/s13075-018-1519-x. PMID 29433546
- [Background] Li S, Yu Y, Koehn CD, Zhang Z, Su K. Galectins in the Pathogenesis of Rheumatoid Arthritis. J Clin Cell Immunol. 2013 Sep 30;4(5):1000164. doi: 10.4172/2155-9899.1000164. PMID 24416634
- [Background] Xia T, Zheng XF, Qian BH, Fang H, Wang JJ, Zhang LL, Pang YF, Zhang J, Wei XQ, Xia ZF, Zhao DB. Plasma Interleukin-37 Is Elevated in Patients with Rheumatoid Arthritis: Its Correlation with Disease Activity and Th1/Th2/Th17-Related Cytokines. Dis Markers. 2015;2015:795043. doi: 10.1155/2015/795043. Epub 2015 Sep 6. PMID 26435567
- [Background] Zhu C, Anderson AC, Kuchroo VK. TIM-3 and its regulatory role in immune responses. Curr Top Microbiol Immunol. 2011;350:1-15. doi: 10.1007/82_2010_84. PMID 20700701
- [Background] Zhu C, Anderson AC, Schubart A, Xiong H, Imitola J, Khoury SJ, Zheng XX, Strom TB, Kuchroo VK. The Tim-3 ligand galectin-9 negatively regulates T helper type 1 immunity. Nat Immunol. 2005 Dec;6(12):1245-52. doi: 10.1038/ni1271. Epub 2005 Nov 13. PMID 16286920